CLINICAL TRIAL: NCT01620983
Title: Knee Arthroplasty Pain Coping Skills Training (KASTPain): A Randomized Trial
Acronym: KASTPain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM14326; 1UM1AR062800-01 (NIH)
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Knee Osteoarthritis
Keywords: arthroplasty; pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pain Coping Skills Training (Experimental): The pain coping skills training will be delivered by physical therapists in eight one-hour sessions by telephone over a 2-month perioperative period. Patients will be taught a variety of skills designed to improve maladaptive pain related thoughts and actions to enhance recovery following arthroplasty.
  Interventions: Behavioral: Pain Coping Skills Training
- Arthritis Education (Active Comparator): The eight one-hour perioperative arthritis education sessions will be delivered by nurse educators via telephone and will use a presentation and discussion format. Figures and discussion sessions will present information on the nature of arthritis, what to expect following knee arthroplasty, treatment of osteoarthritis, the role of exercise, joint protection and making future treatment decisions.
  Interventions: Behavioral: Arthritis Education
- Usual Care (Other): Patients randomly assigned to this arm will undergo usual care following knee arthroplasty.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Pain Coping Skills Training
  Arms: Pain Coping Skills Training
Behavioral: Arthritis Education
  Arms: Arthritis Education
Other: Usual Care
  Arms: Usual Care

SUMMARY:
Patients undergoing knee replacement surgery and who have high levels of pain catastrophizing are at risk for poor outcome. The clinical trial is designed to determine if a pain coping skills training intervention delivered by physical therapists and supervised by psychologists is more effective at reducing pain and improving function and is more cost effective than arthritis education or usual care.

DETAILED DESCRIPTION:
Approximately 25% of patients following knee arthroplasty have disabling pain following apparently successful surgery. Recent research suggests that pain catastrophizing plays a key role in determining which patients with knee arthroplasty have a poor outcome. In addition to this evidence, a substantial literature suggests that pain coping skills training is effective for patients with chronic pain but the intervention has not been studied for surgical patients with severe arthritic knee pain. We designed the Knee Arthroplasty pain coping Skills Training (KASTPain) trial to address this research need. This Phase III three-arm randomized clinical trial seeks to combine a strong and diverse group of researchers to examine an important and understudied area in the joint arthroplasty literature. The KASTPain trial will be the first to examine the utility of a perioperative pain coping intervention for this substantial population of patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults 45 years and older and capable of providing informed consent
* Diagnosis of osteoarthritis as determined by participating orthopaedic surgeons
* Scheduled for an elective unilateral total or unicompartmental knee arthroplasty no sooner than 1 week and no later than 8 weeks from the time of recruitment
* Score of greater than or = to 16 on the Pain Catastrophizing Scale
* Score of greater than or = to 5 on the WOMAC Pain Scale
* Able to read and speak English

Exclusion Criteria:

* Scheduled for revision arthroplasty surgery
* Underwent contralateral knee arthroplasty surgery or hip arthroplasty surgery within 6 months of currently planned surgery
* Unable to or declines study participation
* Self-reported diagnosis of rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosis, ankylosing spondylitis
* Arthroplasty surgery scheduled because of fracture, malignancy or infection
* Scheduled for bilateral arthroplasty surgery
* Scheduled to undergo hip or knee arthroplasty within 6 months of current knee arthroplasty
* Score of 20 or greater on the PHQ-8 depression scale
* Score of less than 3 on the six-item cognitive screener

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2012-12; Primary Completion 2017-06-27 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel L. Riddle, Ph.D., PT, Principal Investigator — Virginia Commonwealth University
Locations (5):
- United States (5):
  - Southern Illinois University, Springfield, Illinois
  - New York University, New York, New York
  - Duke University, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of the main trial, after de-identification.
Supporting Information: Study Protocol
Time Frame: Two years after publication of the primary findings to allow the investigators to publish secondary work from the trial. Data will no longer be available 5 years after publication of the primary findings.
Access Criteria: Proposals must be submitted to the primary investigator who, along with the co-investigators will review the proposal. Access to the dataset will be granted based on scientific merit of the project, absence of overlap with other projects, and impact of the request on other planned uses of the dataset. A signed data user agreement will be required.

REFERENCES:
- [Background] Riddle DL, Keefe FJ, Nay WT, McKee D, Attarian DE, Jensen MP. Pain coping skills training for patients with elevated pain catastrophizing who are scheduled for knee arthroplasty: a quasi-experimental study. Arch Phys Med Rehabil. 2011 Jun;92(6):859-65. doi: 10.1016/j.apmr.2011.01.003. Epub 2011 Apr 29. PMID 21530943
- [Background] Riddle DL, Johnson RE, Jensen MP, Keefe FJ, Kroenke K, Bair MJ, Ang DC. The Pragmatic-Explanatory Continuum Indicator Summary (PRECIS) instrument was useful for refining a randomized trial design: experiences from an investigative team. J Clin Epidemiol. 2010 Nov;63(11):1271-5. doi: 10.1016/j.jclinepi.2010.03.006. Epub 2010 Jun 17. PMID 20670911
- [Background] Riddle DL, Jensen MP, Ang D, Slover J, Perera R, Dumenci L. Do Pain Coping and Pain Beliefs Associate With Outcome Measures Before Knee Arthroplasty in Patients Who Catastrophize About Pain? A Cross-sectional Analysis From a Randomized Clinical Trial. Clin Orthop Relat Res. 2018 Apr;476(4):778-786. doi: 10.1007/s11999.0000000000000001. PMID 29543659
- [Background] Riddle DL, Slover J, Ang D, Perera RA, Dumenci L. Construct validation and correlates of preoperative expectations of postsurgical recovery in persons undergoing knee replacement: baseline findings from a randomized clinical trial. Health Qual Life Outcomes. 2017 Dec 1;15(1):232. doi: 10.1186/s12955-017-0810-x. PMID 29191188
- [Background] Riddle DL, Keefe FJ, Ang D, J K, Dumenci L, Jensen MP, Bair MJ, Reed SD, Kroenke K. A phase III randomized three-arm trial of physical therapist delivered pain coping skills training for patients with total knee arthroplasty: the KASTPain protocol. BMC Musculoskelet Disord. 2012 Aug 20;13:149. doi: 10.1186/1471-2474-13-149. PMID 22906061
- [Derived] Orndahl CM, Perera RA, Riddle DL. Associations Between Physical Therapy Visits and Pain and Physical Function After Knee Arthroplasty: A Cross-Lagged Panel Analysis of People Who Catastrophize About Pain Prior to Surgery. Phys Ther. 2021 Jan 4;101(1):pzaa182. doi: 10.1093/ptj/pzaa182. PMID 32990311
- [Derived] Riddle DL, Slover J, Keefe FJ, Ang DC, Dumenci L, Perera RA. Racial Differences in Pain and Function Following Knee Arthroplasty: A Secondary Analysis From a Multicenter Randomized Clinical Trial. Arthritis Care Res (Hoboken). 2021 Jun;73(6):810-817. doi: 10.1002/acr.24177. PMID 32144884

RESULTS

PARTICIPANT FLOW:
Groups:
- Pain Coping Skills Training: The pain coping skills training will be delivered by physical therapists in eight one-hour sessions by telephone over a 2-month perioperative period. Patients will be taught a variety of skills designed to improve maladaptive pain related thoughts and actions to enhance recovery following arthroplasty.
  Pain Coping Skills Training
- Arthritis Education: The eight one-hour perioperative arthritis education sessions will be delivered by nurse educators via telephone and will use a presentation and discussion format. Figures and discussion sessions will present information on the nature of arthritis, what to expect following knee arthroplasty, treatment of osteoarthritis, the role of exercise, joint protection and making future treatment decisions.
  Arthritis Education
- Usual Care: Patients randomly assigned to this arm will undergo usual care following knee arthroplasty.
  Usual Care
Period: Overall Study
Arm/Group | Pain Coping Skills Training | Arthritis Education | Usual Care
Started | 130 | 135 | 137
Completed | 111 | 113 | 122
Not Completed | 19 | 22 | 15
Not completed — Lost to Follow-up | 8 | 4 | 9
Not completed — Withdrawal by Subject | 6 | 8 | 1
Not completed — Death | 2 | 0 | 0
Not completed — Physician Decision | 3 | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pain Coping Skills Training | Arthritis Education | Usual Care | Total
Number analyzed (Participants) | 130 | 135 | 137 | 402
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (7.9) | 64.2 (8.5) | 62.7 (7.7) | 63.2 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 85 | 88 | 267
  Male | 36 | 50 | 49 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 5 | 13
  Not Hispanic or Latino | 127 | 126 | 130 | 383
  Unknown or Not Reported | 0 | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 4 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 48 | 44 | 47 | 139
  White | 78 | 83 | 86 | 247
  More than one race | 2 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 3 | 1 | 4
WOMAC Pain Scale [Mean (Standard Deviation); unit: units on scale] — A self report scale that quantifies the extent of function limiting pain. The scale ranges from 0 to 20 with higher scores denoting worse activity related pain.
  units on scale | 11.6 (3.1) | 11.3 (3.5) | 11.4 (3.4) | 11.4 (3.4)
WOMAC Function Scale [Mean (Standard Deviation); unit: units on scale] — A self report scale that quantifies the extent of difficulty with daily function. The scale ranges from 0 to 68 with higher scores denoting more difficult daily function.
  units on scale | 38.6 (11.8) | 37.1 (11.8) | 36.0 (11.1) | 37.2 (11.6)
Pain Catastrophizing Scale [Mean (Standard Deviation); unit: units on scale] — A scale that quantifies the extent to which a participant catastrophizes about their pain. Score range from 0 to 52 with higher scores denoting greater pain catastrophizing
  units on scale | 30.4 (9.6) | 30.0 (9.2) | 29.7 (9.2) | 30.0 (9.3)
Six minute walk test [Mean (Standard Deviation); unit: meters] | 305 (121) | 279 (132) | 309 (106) | 297 (120)
Short Physical Performance Battery [Mean (Standard Deviation); unit: units on scale] — The Short Physical Performance Battery measures actual physical performance of four common daily physical activities including standing balance, single standing from a chair, repeated standing from a chair, and a 4 meter walk test. Scores range from 0 to 12 with higher scores indicating better physical performance.
  units on scale | 7.6 (3.2) | 7.5 (2.9) | 7.9 (2.6) | 7.8 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Scale
Description: A self report scale that quantifies the extent of function limiting pain. The scale ranges from 0 to 20 with higher scores denoting worse activity related pain.
Time Frame: twelve months
Population: Data from all subjects were included in primary and secondary analyses.
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Pain Coping Skills Training | Arthritis Education | Usual Care
Number analyzed (Participants) | 130 | 135 | 137
units on scale | 3.3 [2.5 to 4.2] | 3.0 [2.1 to 3.8] | 2.9 [2.0 to 3.8]

2. Secondary Outcome: WOMAC Physical Function Scale
Description: A self report scale that quantifies the extent of difficulty with everyday activity. The scale ranges from 0 to 68 with higher scores denoting greater difficulty with daily function.
Time Frame: twelve months
Population: Data from all subjects were included in the analyses.
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Pain Coping Skills Training | Arthritis Education | Usual Care
Number analyzed (Participants) | 130 | 135 | 137
units on scale | 12.2 [9.0 to 15.4] | 11.7 [8.6 to 14.9] | 10.5 [7.4 to 13.6]

3. Secondary Outcome: 0 to 10 Verbal Pain Rating Scale
Description: An 11 point verbal pain rating scale with higher scores denoting higher pain intensity.
Time Frame: twelve months
Population: Data from all subjects were included in the analyses.
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Pain Coping Skills Training | Arthritis Education | Usual Care
Number analyzed (Participants) | 130 | 135 | 137
units on scale | 1.8 [1.2 to 2.4] | 2.0 [1.3 to 2.6] | 1.7 [1.1 to 2.2]

4. Secondary Outcome: Pain Catastrophizing Scale
Description: A scale that quantifies the extent to which a participant catastrophizes about their pain. Score range from 0 to 52 with higher scores denoting greater pain catastrophizing.
Time Frame: twelve months
Population: Data from all subjects were included in the analyses.
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Pain Coping Skills Training | Arthritis Education | Usual Care
Number analyzed (Participants) | 130 | 135 | 137
units on scale | 6.8 [4.0 to 9.6] | 7.2 [4.0 to 10.0] | 6.1 [3.4 to 8.9]

5. Secondary Outcome: Global Rating of Change Scale
Description: 11 point scale ranging from -5 to +5 with higher scores denoting a greater recovery.
Time Frame: twelve months
Population: Data from all subjects were analysed.
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Pain Coping Skills Training | Arthritis Education | Usual Care
Number analyzed (Participants) | 130 | 135 | 137
units on scale | 3.6 [3.1 to 4.2] | 3.8 [3.3 to 4.3] | 4.1 [3.6 to 4.6]

6. Secondary Outcome: Six-minute Walk Test
Description: Distance walked in six minutes.
Time Frame: twelve months
Population: Data from all subjects were analysed.
Measure: Mean (95% Confidence Interval); unit: meters
Arm/Group | Pain Coping Skills Training | Arthritis Education | Usual Care
Number analyzed (Participants) | 130 | 135 | 137
meters | 366 [341 to 391] | 337 [313 to 362] | 363 [340 to 387]

7. Secondary Outcome: Short Physical Performance Battery
Description: The Short Physical Performance Battery measures actual physical performance of four common daily physical activities including standing balance, single standing from a chair, repeated standing from a chair, and a 4 meter walk test. Scores range from 0 to 12 with higher scores indicating better physical performance.
Time Frame: twelve months
Population: Data from all subjects were analysed.
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Pain Coping Skills Training | Arthritis Education | Usual Care
Number analyzed (Participants) | 130 | 135 | 137
units on scale | 8.4 [7.6 to 9.1] | 8.0 [7.2 to 8.7] | 8.8 [7.8 to 9.4]

ADVERSE EVENTS:
Time Frame: Adverse events were collected both from the participants, and from the medical record over the time period from the time of surgery to 12 months following surgery.
Description: The time frame has not changed from the original definition. The sample size for persons experience adverse events or serious adverse events is different from baseline consent because 18 subjects who consented to participate did not have knee replacement surgery and therefore were not considered for adverse events.Of the 18, 5 were randomly assigned to the usual care arm at baseline, 10 were assigned to the arthritis education arm and 3 were assigned to the pain coping skills training arm.
Arm/Group | Pain Coping Skills Training | Arthritis Education | Usual Care
All-Cause Mortality (participants affected / at risk) | 2/127 | 0/125 | 0/132
Serious Adverse Events (participants affected / at risk) | 34/127 | 36/125 | 28/132
Other Adverse Events (participants affected / at risk) | 8/127 | 3/125 | 9/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pain Coping Skills Training (N=127) | Arthritis Education (N=125) | Usual Care (N=132)
venous thromboembolism (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 3 (3)
infection of knee (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2)
Hospitlilization (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 5 (5) — Other hospitalization other than the index knee
Hospitalization for psychological distress (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Revision of index knee (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 1 (1)
Manipulation of index knee (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (7) | 3 (3) — Due to stiffness
Contralateral knee replacement (Musculoskeletal and connective tissue disorders) | 12 (12) | 13 (13) | 7 (7)
Other hospitalization (Surgical and medical procedures) | 7 (7) | 7 (7) | 7 (7) — Non-musculoskeletal admissions
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pain Coping Skills Training (N=127) | Arthritis Education (N=125) | Usual Care (N=132)
psychological distress (Nervous system disorders) | 5 (5) | 2 (2) | 8 (8)
shortness of breath (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
orthopaedic injury to the knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Emergency room visity for knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
No limitations were noted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-07-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT01620983/Prot_SAP_000.pdf